CLINICAL TRIAL: NCT04452617
Title: Safety of Short-term Hydroxychloroquine Plus Azithromycin Treatment in Critically Ill Patients With Severe COVID-19
Status: Completed | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: REA-03-2020
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: hydroxychloroquine; ADRS; azithromycine; torsade de pointe
MeSH Terms: conditions — COVID-19; Torsades de Pointes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hydroxychloroquine and azithromycin have been proposed as treatment of COVID-19 patients, but few reports have assessed this combination therapy in critically ill COVID-19 patients.

Many raised concerns regarding the potential cardiac toxicity of this association.

The purpose of this monocenter retrospective observational study is to evaluate the safety of a short term treatment with hydroxychloroquine and azithromycin in critically ill patients admitted in ICU for severe COVID-19 with respiratory failure.

The main objective is to assess the incidence of severe cardiac arrhythmia e.g torsade de pointes and cardiac arrest or sudden death, during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients admitted in ICU for severe COVID-19 with respiratory failure for at least two days of treatment with hydroxychloroquine and azithromycin.

Exclusion Criteria:

* cardiac conduction disorders
* continuous anti-arrhythmic therapy
* heart failure
* chronic renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted in ICU for severe COVID-19 with respiratory failure and a short term treatment with hydroxychloroquine (HCQ) and azithromycin (AZ):
  * HCQ administered at a daily dosage of 600mg in 3 doses for 10 days.
  * AZ administered at a dosage of 500mg on the first day and then 250mg/day for 4 to 6 days.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
occurrence of severe cardiac arrhythmia: torsade de pointes and cardiac arrest or sudden death | 30 days after admission in ICU

SECONDARY OUTCOMES:
assessment of QTc interval prolongation during the treatment period compared to baseline ECG | daily
  QTc (corrected QT interval) > 500 ms and ΔQTc > 60 ms

CONTACTS AND LOCATIONS:
Overall Officials: Lyes KNANI, Doctor, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No